CLINICAL TRIAL: NCT03477487
Title: Preliminary Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Osteoarthritic Pain
Brief Title: Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Osteoarthritic Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xalud Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XT-150-1-0202
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis, Knee
Keywords: inflammation; Cytokines; Interleukin-10; Gene therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation

STUDY DESIGN:
Intervention Model Description: Ascending dose-ranging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lowest dose (Experimental): The lowest dose of XT-150 in the escalation schedule
  Interventions: Biological: XT-150
- Second dose (Experimental): The 2nd dose of XT-150 in the escalation sequence
  Interventions: Biological: XT-150
- Third dose (Experimental): The 3rd dose of XT-150 in the escalation sequence
  Interventions: Biological: XT-150
- Highest dose (Experimental): The highest dose of XT-150 in the escalation sequence
  Interventions: Biological: XT-150

INTERVENTIONS:
Biological: XT-150 — Human IL-10 variant transgene in a plasmid DNA vector

SUMMARY:
Evaluation of Safety, Tolerability, and Efficacy of XT-150, a plasmid DNA with a variant of human IL-10 transgene. XT-150 will be a single injection into the knee synovial capsule for the Treatment of Osteoarthritic Pain.

DETAILED DESCRIPTION:
Phase 1 dose escalation study to evaluate the safety, tolerability, and efficacy of a plasmid DNA encoding a variant of human IL-10. This 6-month study will follow subjects with severe osteoarthritis of the knee. Safety labs, physical exams, and blood levels of the IL-10 variant will be assessed for tolerability and any adverse events associated with the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 90 years of age, inclusive
2. Sufficiently severe OA of the knee to meet accepted criteria for knee arthroplasty
3. Free of intra-articular infection, or infection at the injection site.
4. Symptomatic disease because of osteoarthritis, defined as one or more of the following Visual Analog Scale of Pain Intensity (VASPI) scores:

   1. a worst pain of at least 70 at any time during the preceding week (based on scale of 0 to 100, with 100 representing "pain as bad as you can imagine").
   2. a worst stiffness of at least 70 at any time during the preceding week (based on a scale of 0 to 100, with 100 representing "stiffness as bad as you can imagine").
5. Stable analgesic regimen during the 4 weeks prior to enrollment.
6. Inadequate pain relief (minimum ≥5 mean on the Brief Pain Inventory-Severity Scale) lasting ≥3 months.
7. In the judgment of the Investigator, acceptable general medical condition
8. Life expectancy >6 months
9. Female subjects of child-bearing potential, and those <1 year post-menopausal, must be practicing effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm) or total abstinence from heterosexual intercourse for a minimum of 1 month before study drug administration and agree to continue prevention methods for 3 months after participation in the study is completed.
10. Male subjects who are heterosexually active and not surgically sterile must agree to use effective contraception, including abstinence, for the duration of the study and for 3 months after the study is completed.
11. Have suitable knee joint anatomy for intra-articular injection
12. Willing and able to return for the follow-up (FU) visits
13. Able to reliably provide pain assessment
14. Able to read and understand study instructions, and willing and able to comply with all study procedures

Exclusion Criteria:

1. 1. Hypersensitivity, allergy, or significant reaction to any ingredient of the study drug, including double-stranded DNA, mannose, and sucrose
2. Subject plans knee arthroplasty within 4 months, irrespective of the outcome of the trial or other conservative therapies
3. High peri-procedural risks which in the judgment of the investigator preclude a safe knee injection procedure (e.g., poorly controlled diabetes, cardiac inadequacy such as NYHA class > II, G4 glomerular filtration rate [eGFR < 30 mL/min by Cockcroft-Gault])
4. Current treatment with immunosuppressives (steroid therapy equivalent to >10mg/day prednisone); or other strong immunosuppressant
5. History of systemic immunosuppressive therapy; steroids (equivalent to >10mg/day prednisone) in the last 3 months
6. Currently receiving systemic chemotherapy or radiation therapy for malignancy
7. Clinically significant hepatic disease as indicated by clinical laboratory results ≥3 times the upper limit of normal for any liver function test (e.g., aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase)
8. Severe anemia (Grade 3; hemoglobin <8.0 g/dL, <4.9 mmol/L, <80 g/L; transfusion indicated), uncontrolled coagulopathy (Grade 1, prolonged activated partial prothrombin time (aPTT) > upper limit of normal (ULN) to 1.5xULN), or bleeding diathesis, Grade 1 white cell counts (lymphocytes <LLN - 800/mm3; <LLN - 0.8 x 10e9 /L, neutrophils <LLN - 1500/mm3; <LLN - 1.5 x 10e9 /L)
9. Positive serology for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus within 4 weeks of commencing the study
10. Significant neuropsychiatric conditions; dementia, major depression, or altered mental state that in the opinion of the Investigator will interfere with study participation
11. Current treatment with systemic antibiotics or antivirals (EXCEPTION: topical treatments)
12. Current treatment with anticoagulants, other than low-dose aspirin, prescribed for new onset of symptoms in 3 months before screening visit.
13. Known or suspected history of active alcohol or intravenous/oral drug abuse within 1 year before the screening visit
14. Women who are pregnant or nursing
15. Use of any investigational drug or device within 1 month before enrollment or current participation in a trial that included intervention with a drug or device; or currently participating in an investigational drug or device study.
16. Any condition that, in the opinion of the Principal Investigator, could compromise the safety of the subject, the subject's ability to communicate with the study staff, or the quality of the data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months
  Clinical, laboratory measures of safety by CTCAE v4.0

SECONDARY OUTCOMES:
Visual Analog Scale of Pain Intensity | 6 months
  Validated index of pain
Knee Injury and Osteoarthritis Outcomes Scale | 6 months
  KOOS
WOMAC | 6 Months
  Western Ontario and McMasters University Osteoarthritis Index
Brief Pain Inventory | 6 months
  Measure of pain associated with osteoarthritis

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Collins, MD, PhD, Study Director — Xalud Therapeutics, Inc.
Locations (1):
- Neurovations (Napa Pain Institute), Napa, California, United States

IPD SHARING:
Plan to Share IPD: No